CLINICAL TRIAL: NCT01166152
Title: Development of a New Diagnosis and Intervention Method for Developmental Disorders
Acronym: DIDD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tokyo University of Agriculture and Technology (Other)
Collaborators: Ashiya University (Other); Saitama Medical University (Other)
Responsible Party: Shun Nakamura/Professor, Tokyo University of Agriculture and Technology
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: TokyoUAT_21_11
Record Dates: First submitted 2010-07-19; First posted 2010-07-20 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2010-07

CONDITIONS: Developmental Disabilities
Keywords: autistic spectrum disorders; developmental disorders
MeSH Terms: conditions — Developmental Disabilities; Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Behavioral: social skills training — meeting once a week or biweekly to play together using toys, games, and physical exercises.

SUMMARY:
The purpose of this study is to develop a new diagnostic method for developmental disorders based on behavior recording during the interview of the subjects by medical staff as well anonymous persons. The behavior recording by video camera will be accompanied by non-invasive physiological recordings, including electroencephalogram (EEG), electrocardiogram (ECG), electromyogram (EMG), and body temperature using infrared (IR) thermograph. Thus, the physiologically relevant and the disorder correlated behavior parameters could be extracted and used as new diagnostic markers. If necessary, the medical staff may take blood sample from the subject before and after the interview. For the longitudinal study, the similar interview and the recording of the same subject will be planned to evaluate the effect of the medical and educational intervention. The investigators also examine the synergistic effect of the intervention and the administration of the supplement (e.g., vitamin D, arachidonic acid, coenzyme Q10 (CoQ-10)). The clinician may use Risperidone.

DETAILED DESCRIPTION:
Case 1:The investigators started the intervention and supplementation of arachidonic acid for 3 patients diagnosed as autistic spectrum disorders (ASD) from September 4, 2010 at Sawa hospital (Osaka, Japan). Another ASD patients (n=5) at Sawa hospital were treated by administration of Risperidone as medicinal drink from January 14, 2011. The supplementation as well as Risperidone administration followed double-blind placebo controlled cross-over protocol to access the effect of the treatment. These trials will continue until November 2011. Final outcome will be evaluated by clinical diagnosis and behavior parameters measurement as described under Brief Summary.

Case 2: The investigators started the intervention and supplementation of reduced form of CoQ10 for learning disability children (n=20) at small private cramming school (JIZAI-ken, Tokyo) from February 5, 2011. This trial will continue until October 2011. The effect of the intervention and supplementation will be evaluated by behavior parameter measurement as described above.

ELIGIBILITY:
Inclusion Criteria:

* Developmental disorders

Exclusion Criteria:

* Mental retardation

Max Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-08; Primary Completion 2011-11 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
thermogram of head | at least 8 weeks after intervention
  The themogram of head will be measured using IR camera (TVS-500EX, NEC Avio) during clinical interview to see the change of autonomic nervous system activity.

SECONDARY OUTCOMES:
view direction | at least 8 weeks after intervention
  The subject view direction will be monitored using the video camera (Sony) during clinical interview.

CONTACTS AND LOCATIONS:
Overall Officials: Kunio Yui, MD, PhD, Principal Investigator — Ashiya University; Hideo Yamauchi, MD, PhD, Principal Investigator — Saitama Medical University; Mamiko Koshiba, PhD, Principal Investigator — Tokyo University of Agriculture and Techinology; Shun Nakamura, PhD, Principal Investigator — Tokyo University of Agriculture and Techinology
Locations (1):
- Ashiya University Graduate School of Clinical Education, Ashiya, Hyōgo, Japan